CLINICAL TRIAL: NCT07249021
Title: Integration of Multi-modality Imaging Protocols With emphAsis on CT in Image Guided Adaptive Brachytherapy (IGABT) for Cervical Cancer - EMBRACE III-IMPACT STUDY
Brief Title: This is a Multicentre International Study Evaluating CT-based IGABT With / Without Either TRUS During BT/Pre BT MR as Per IBS-GECESTRO-ABS Recommendations for Target contouring-as an Alternative to MRIGABT for Cervical Cancer From Implementation Perspectives Under EMBRACE-III:TRIPLET IMPACT Study.
Acronym: IMPACT
Status: Not yet recruiting | Type: Observational
Sponsor: Homi Bhabha Cancer Hospital & Research Centre (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Umesh Mahantshetty, Professor, Homi Bhabha Cancer Hospital & Research Centre
Other Study IDs: IEC/0725/12000090/001
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Cervical Cancer; Brachytherapy; CT; Transrectal Ultrasound
Keywords: Cervical cancer; CT-guided brachytherapy; Image-Guided Adaptive Brachytherapy (IGABT); Locally advanced cervical cancer; Implementation study; Resource-limited settings; Low- and middle-income countries (LMICs); EMBRACE III; Trans-rectal ultrasound during BT; Pre BT MR Imaging
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort A - Advanced CT Environment, Cohort B - Basic CT Environment: COHORT A: Pre Brachytherapy MR to assess the regression of primary tumour after EBRT +/- CT, defining target and pre-planning of BT implantation followed by CT Imaging with BT applicator in place. Alternatively, if Pre-BT MR is not feasible, use of TRUS imaging information during BT application to define the target on CT Imaging with BT applicator in situ
  COHORT B: CT Imaging with BT Applicator in place-based treatment planning for each BT application.
  Interventions: Other: CT IGABT

INTERVENTIONS:
Other: CT IGABT — Participants with locally advanced cervical cancer will receive standard-of-care treatment, including external beam radiotherapy (EBRT) with concurrent weekly cisplatin chemotherapy, followed by image-guided adaptive brachytherapy (IGABT). Brachytherapy planning will utilize CT-based imaging to define target volumes and organs at risk according to international consensus guidelines. Centres with advanced imaging capabilities may integrate MRI or transrectal ultrasound (TRUS) for pre-brachytherapy assessment (Cohort A), while others will use CT-only planning (Cohort B). All treatments will follow standardized protocols with centralized quality assurance and data review to evaluate feasibility, consistency, and clinical outcomes of CT-IGABT implementation across diverse clinical environments.

SUMMARY:
Title: Integration of Multi-modality Imaging Protocols with Emphasis on CT in Image-Guided Adaptive Brachytherapy (IGABT) for Cervical Cancer - EMBRACE III-TRIPLET : IMPACT Study Locally advanced cervical cancer (LACC) remains a major health challenge, particularly in low- and middle-income countries (LMICs), which account for the majority of global cases. The standard curative treatment involves a combination of external beam radiotherapy (EBRT) with concurrent chemotherapy, followed by brachytherapy (BT). Brachytherapy plays a crucial role in achieving high local control by delivering radiation directly to the tumour through internally placed radioactive sources.

Historically, BT dose prescription was based on two-dimensional (2D) X-ray images and defined anatomical "points," achieving 5-year local control rates of 60-70%. Over the last decade, magnetic resonance imaging (MRI)-based image-guided adaptive brachytherapy (MR-IGABT) has transformed practice by enabling three-dimensional (3D) target-based dose prescription and adaptation to tumour regression. The landmark EMBRACE I study, involving over 1300 patients, demonstrated over 90% 5-year local control rates with MR-IGABT, establishing it as the international gold standard endorsed by NCG, ICRU, NCCN, and ESGO-ESTRO guidelines.

However, MRI-based planning for IGABT remains logistically and financially challenging for many centres, especially in LMICs. CT and transrectal ultrasound (TRUS) have emerged as feasible alternatives, offering broader accessibility. Despite encouraging outcomes from smaller institutional studies, the lack of standardized and validated target delineation concepts for CT-IGABT has led to significant variability in clinical implementation. Recognizing this, the Indian Brachytherapy Society (IBS), American Brachytherapy Society (ABS), and GEC-ESTRO jointly published consensus recommendations in 2020 to standardize CT-IGABT practices across diverse clinical environments.

At Homi Bhabha Cancer Hospital and Research Centre, Visakhapatnam, our prior work (RetroLACER Study) demonstrated that CT-based IGABT can achieve outcomes comparable to MR-IGABT, highlighting its feasibility and potential for wider adoption. Building on this foundation, the EMBRACE III-IMPACT Study seeks to evaluate whether CT-IGABT can be systematically and uniformly implemented in a multi-centre setting and to benchmark clinical outcomes against the standards set by MR-IGABT.

Study Design:

This is a multicentre, prospective, observational study planned to include approximately 1200 participants with locally advanced cervical cancer. All participants will receive standard-of-care treatment, including EBRT, concurrent weekly cisplatin chemotherapy, and brachytherapy with image-guided planning.

Objectives:

To assess the feasibility of implementing standardized CT-IGABT protocols across diverse clinical environments.

To evaluate local control, disease-free survival, and treatment-related toxicity outcomes for CT-IGABT.

To compare and benchmark CT-IGABT outcomes with established MR-IGABT benchmarks from prior international studies.

Participant Involvement:

Participants will undergo standard diagnostic imaging, EBRT with weekly cisplatin, and brachytherapy using CT-based planning. Imaging and treatment data will be collected, anonymized, and submitted to a central database for review. Regular follow-up visits will monitor tumour control and treatment-related side effects.

Benefits:

Participants receive internationally standardized, quality-assured treatment protocols. Centres gain access to expert review and QA support from international collaborators, potentially improving treatment quality and outcomes.

The study supports global efforts to establish CT-IGABT as a cost-effective, accessible alternative to MRI-based IGABT, expanding equitable cancer care access.

Risks:

The study is observational and involves standard treatment; therefore, risks and costs are comparable to routine cervical cancer care.

Confidentiality and Ethics:

All data will be anonymized and handled in compliance with ethical and regulatory standards. Participant confidentiality will be strictly maintained. Written informed consent will be obtained before study participation.

Significance:

By validating standardised CT-based protocols and establishing outcome benchmarks, the study aims to facilitate widespread adoption of IGABT in resource-limited settings, ultimately improving treatment accessibility and survival outcomes.

DETAILED DESCRIPTION:
The study is a multi-centre prospective observational study. Reporting on the key clinical treatment and outcome parameters are mandatory for the individual centre.

The study will evaluate CT-IGABT for cervical cancer in two different CT based clinico- radiological environments.

Cohort A - Advanced CT Environment: [CT or MR at Diagnosis] and [ (Pre BT MR or TRUS) and CT at BT] Cohort B - Basic CT Environment: [CT or MR at Diagnosis] and [CT at BT]

After satisfying the inclusion and exclusion criteria, patients will be taken up in the study.

External Beam Radiotherapy:

The primary focus of this protocol is to prospectively validate the target volume concepts and benchmark the clinical outcomes with CT based IGABT for cervical cancer. However, for the overall outcome of the study with regards to secondary endpoints like regional control and survival as well as to morbidity, the contribution from EBRT may have a certain impact. Harmonization of dose and volume components of EBRT for targets (local and regional) as well as organs at risk is mandatory to ensure comparable treatment volumes across treating centres. Nomenclature of targets and organs at risk preferably needs to be uniform and in line with the EBRT protocols of EMBRACE-II study to maintain uniform reporting. Contrast CT scan in supine position with adequate positioning and immobilisation as per institutional protocols is mandatory for planning, with a slice thickness not exceeding 5 mm (preferably 1-3 mm). Oral contrast and vaginal markers are optional, as per institutional protocols. A reproducible protocol for bladder and rectal filling (at the time of simulation as well as treatment delivery) is mandatory and may be adopted as per institutional protocols. Delineation of target volumes and organs at risk should be done on the planning CT scan, taking into consideration all the information obtained from diagnostic and staging investigations including clinical drawings and NMD's. CTV_T should include the cervix, parametrium, entire uterus (and adnexa), and 2cm of uninvolved vagina as a minimum. Involved lymph nodes should be contoured as GTV_N and an optional margin of 0 to 3mm may be given to generate CTV_N. Lymph nodal regions to be included in elective nodal CTV (CTV_E). ITV and PTV should be generated around the CTV_T as per institutional practice (population based generic margins, or patient specific margins based on empty and full bladder scans) and should reflect the protocol employed for reproducible bladder and rectal filling. In general, a total safety margin of approximately 1 to 1.5cm is recommended around the CTV_T (including ITV and PTV). A PTV should be generated around CTV_E, and CTV_N as per institutional practice for elective and involved nodal boost volumes, respectively.

For uniform reporting of EBRT dose-volume parameters, the final PTVs should be labelled as PTV_Prescribed Dose (Eg: PTV_45, PTV_55, etc).

The dose contribution from EBRT must be homogenous for patients included in this study, especially in regions corresponding to the small volumes of interest for BT (CTV-THR-CT and adjacent OARs like anterior-lateral walls of rectum and sigmoid, posterior-inferior wall of the bladder, walls of the vagina adjacent to macroscopic disease, etc). Such homogeneity ensures optimal comparison of dose-volume effects of BT on local control and morbidity.

For reporting dose in defined absolute tissue volumes it is necessary to report the dose for EBRT in each OAR. It is assumed that the small volumes of interest for BT will receive the EBRT dose prescribed to PTV. Therefore, no additional dose volume assessment is required for the different organs at risk, apart from the confirmation that the EBRT dose received in the volumes of interest does not exceed the prescribed dose by ± 5%. If nodal boost given by EBRT is contributing to a specific OAR volume adjacent to / overlapping with the target of interest for BT, the total dose including the EBRT boost dose received by that organ must be reported and used for the cumulative EQD2 calculations for that OAR. Dose volume constraints being utilized in the EMBRACE II protocol may be used as a general reference for treatment planning (Annexure-5). Participating institution to evaluate their EBRT plans, especially when IG-IMRT and/or simultaneous integrated boost techniques are used.

Physical dose ranges for EBRT should not be beyond the range of 45 to 50 Gy in conventional fractionation of 1.8 to 2 Gy per fraction and 5 fractions a week. To compensate for unplanned treatment breaks, however, two daily EBRT fractions at least 6 hours apart may be used. To minimize the risk of consequential late damage, dose accumulation of EBRT must, however, not exceed 12 Gy per week. A nodal boost equivalent to a cumulative dose of 55 to 60 Gy (10) (including potential contribution from BT) may be used for node positive disease, as per institutional practice. Nodal boost may be delivered either as simultaneous integrated boost (SIB) or sequential boost (SEB) using IG-IMRT, without compromising on the overall treatment time. Parametrial / nodal EBRT boost through midline shielding or 3D-CRT is not allowed.

Based on the observations from EMBRACE I study, overall treatment time (OTT) has a significant impact on local control probability. Therefore, OTT (including EBRT, BT and concurrent chemotherapy) must be limited to less than 49 days. Any prolongation in OTT beyond 49 days should be documented and reported, along with specific reasons for such prolongation.

Reporting EBRT parameters:

* Dose per fraction, number of fractions, total prescription for each target
* Overall treatment time of whole EBRT
* Dose Volume parameters for EBRT as per CRF

  * Body Absolute volume (in cc) receiving atleast 43 Gy dose (V43Gy )
  * Volume (in cc) of PTV-E

Concomitant chemotherapy:

Cisplatin is to be given intravenously at a dose 40 mg/m2 once a week for a total of preferably 5-6 cycles during the entire course of radiotherapy including BT, according to institutional practice. Patients not suitable for cisplatin chemotherapy are to be excluded from the IMPACT study. Cisplatin dosing may be adjusted / withheld at the discretion of the treating physician, based on tolerance and hematological / renal parametres.

Response to EBRT + Concomitant Chemotherapy:

The categorical classification system is based on the disease extent of the cervix, parametria, vagina, uterine corpus, bladder and rectum at diagnosis and at BT as per IBS-GEC ESTRO - ABS Guidelines.

Brachytherapy:

Treatment planning and performance of BT is based on the recommendations of the "ICRU 89/GEC ESTRO Report" on "Prescribing, Recording and Reporting Brachytherapy for Cancer of the Cervix" (ICRU Report 89, 2013/2016) where the concepts and parameters for image guided adaptive brachytherapy are systematically described.

Overall Schedule for EBRT and BT and chemotherapy:

The overall treatment time (OTT), defined from the first external beam fraction to the end of brachytherapy fraction dose delivered should be < 49 days. This is based on the Retroembrace and Embrace I clinical outcome studies.

To obtain maximal tumour regression the treatment should always be initiated with EBRT and concomitant chemotherapy for 4-5 weeks before BT is applied in weeks 5-7. For a small and/or well responding tumour BT may be initiated already during EBRT to shorten the overall treatment to 5-6 weeks. In any case every effort should be made to keep the overall treatment time < 49 days.

Concomitant chemotherapy given on the first 2-3 days of the week also theoretically paves the way for sensitizing more fractions of EBRT in that week, rather than giving chemotherapy towards the weekend where the sensitizing effect is expected to vanish during the weekend. There is limited data on the optimal timing of EBRT and concomitant chemotherapy on the actual day where it is given. Centres can use their own schedule. Minimum of 5 cycles of cisplatin should be delivered throughout the radiation therapy including BT to ensure optimal outcome from concomitant chemotherapy effect.

Pre-Brachytherapy Planning:

For an ideal brachytherapy application for cervix cancer, a pre-planning procedure is essential which allows tailoring the BT application based on tumour topography and patient anatomy at the time of brachytherapy. This requires a comprehensive clinical gynaecologic examination assessing utero-vaginal topography, tumour response at the primary, parametria and vagina after external beam therapy. Precise documentation on the standard gynaecologic template in three orientations including the speculum view is mandatory. These findings can be supported by volumetric imaging like pre-BT MRI, TRUS imaging during BT application to efficiently define the NMD's on CT with BT applicator in situ. An individual adaptive CTV-THR is defined with a certain width, thickness and height based on the above information. Essential are the correlation of these CTV dimensions to cervical canal, later location of tandem, in particular, distances to outer borders of the contemplated CTV-THR and if symmetrical or not. A calculated decision is taken regarding type of application, in particular, if it can be only intracavitary or a combination of intracavitary and interstitial application. The most precise pre-treatment planning is with a tandem and vaginal applicators in place, and position of needles decided on the image taken according to extent of high- risk CTV. The type of BT application, use of interstitial tubes /needles, pre-BT MR protocol with/without tandem/vaginal applicator for each case is at the discretion of the treating physician and Institutional practice.

Based on the Imaging Environment during BT, two clinical scenarios for CT based BT planning can be utilized. BT treatment with more than 1 BT fraction for every BT application is allowed for either environment.

A. Advanced CT Environment: Pre BT MR to assess the regression of primary tumour after EBRT +/- CT, defining target and pre-planning of BT implantation followed by CT Imaging with BT applicator in place. Alternatively, if Pre-BT MR is not feasible, use of TRUS imaging information during BT application to define the target on CT Imaging with BT applicator in situ.

B. Basic CT Environment: CT Imaging with BT Applicator in place-based treatment planning for each BT application.

Patient preparation for BT Application:

Detailed counselling helps in patient acceptance and compliance to application and treatment. Fitness for anaesthesia will be obtained. In case of co-morbidities, adequate time for optimization of drug regimens is provided without compromise in overall treatment time. The practice of ward admission 1 day prior to BT application is encouraged. Bowel preparation is always to be used to ensure relatively empty recto-sigmoid and small bowel, which is of particular importance when interstitial needles in addition to intracavitary treatment are used and if more than one fraction of BT treatment is planned with same application. This would help to prevent major variations in OAR volumes and subsequently the DVH parameters. Supportive treatment such as DVT prophylaxis (lower limb stockings / low molecular weight heparin), antibiotics and analgesics may be given according to individual patient needs and institutional practice.

BT Applicator Implantation:

The procedure should be performed under anaesthesia (General /spinal) with /without sedation. Strict asepsis throughout the BT procedure has to be maintained. Bladder catheterization with 7 ml of normal saline/ distilled water (high density contrast should be avoided) to inflate the foley's balloon and maintaining the tip end towards base of bladder and a mild negative suction using asepto syringe is recommended.

A thorough clinical assessment under anaesthesia with description of primary tumoral extension, and involvement of parametria, vagina, bladder and rectum are mandatory. In addition, tumour dimensions (width, height and thickness) and clinical NMD (right & left) in relation to central cervical canal is to be noted. Examination findings are documented in clinical drawing sheets. Sounding and dilatation if required of the utero-cervical canal can be guided by trans-abdominal or trans-rectal ultrasound and the length of uterine cavity is measured. Hydrometra / Pyometra (culture and antibiotic sensitivity if required) may be drained if present. A CT/MRI compatible BT applicator is chosen depending on topography of tumour, utero-cervical canal length, vaginal capacity. Choice of applicator type (IC / IC+IS) depends on individual anatomy, clinical NMD's, asymmetry of target topography and tumour spread at the time of brachytherapy. Applicator type (e.g. ring or ovoid type) can be decided by the treating physician. Additional implantation of CT/MR compatible needles/plastic tubes in the parametrium and/or vagina must be used as appropriate for adequate target coverage. Vaginal packing must be performed with gauze (without radio-opaque marker) to push away the rectum and bladder and to fix the applicator against the cervix. The gauze may be soaked with betadine or US gel or saline water to distinguish the packing from vaginal walls.

If TRUS imaging is performed during BT application, a set of images - axial and sagittal are acquired with tandem in place and TRUS based NMD's are measured. Applicator may be fixed to the patient by elastic T shaped bandages. Alternatively, an individual mould or other customized procedures may be used for fixation of applicator as per participating institutional practice. Fixed geometry of applicator in relation to target volume is critical for safe delivery of treatment plan. External fixation to the surgical table/board should not be used. In-vivo dosimetry by use of detectors may be used according to institutional practice. Patient is transferred to CT scanner to obtain appropriate images with the patient in supine treatment position with a specified protocol as detailed below.

Imaging for pre planning and planning to be performed as per environments is as follows:

Imaging Protocols for Brachytherapy:

1. Pre BT MRI:

   MRI, the gold standard, is highly accurate (i) for GTV (high signal intensity zone on T2) assessment including the uterine cervix, parametria, uterine corpus, vagina and for organ wall involvement (bladder, rectum) and (ii) for identifying "grey zones" on T2 in the region of the initial GTV, which are used for the definition of the CTV-THR. Pre BT (preferably within 1 week of EBRT completion) Pelvic MRI should be performed with a well-defined protocol including patient position, use of a pelvic coil, introduction of vaginal ultra- sound gel, bladder and rectal filling protocols and appropriate standard sequences as recommended by GEC -ESTRO. Standardization of protocol prior to implementation is required along with defining an institutional bladder filling protocol. A minimum of T1 (as image localizer) and T2 weighted FRFSE non-contrast, axial, sagittal and coronal (para-axial / para-sagittal or para-coronal) sequences with 3-5 mm slice thickness, 0-2 mm spacing and 256 x 256 matrixes using 0.35 - 3 Tesla MR is preferred.
2. TRUS:

   TRUS has been used to define target structure in relation to cervical canal at the time of BT which corresponds to target structure on MRI. The CTV-THR contains structures which appear dark (hypo- echoic) on ultrasound image: residual GTV, cervical stroma, extra-cervical residual GTV and/or parametrial fibrotic pathologic tissue. There is a significant contrast between normal fatty parametrial tissue (bright) and adjacent pathologic tissue (dark - hypo-echoic) which allows for defining and contouring the target.

   TRUS with biplanar probes and acquisition of images at various levels of cervical canal in relation to uterine vessels, external and internal os, provide useful information to define the target accurately as compared to stand-alone CT images. In-room intraoperative ultrasonography with a trans-rectal (5 - 7.5 MHz) probe can be used to guide and facilitate the application especially placement of uterine tandem to prevent uterine perforations. The TRUS probe is covered with sterile gel inside a plastic sheath and axial images can be acquired transrectally after the placement of tandem into the utero-cervical canal. With the uterine tandem in situ, scanning of cervical region is done to identify uterine arteries (assisted & confirmed by color doppler). From the level of these uterine vessels, a series of trans-axial images in inferior direction can be obtained by retracting TRUS probe sequentially. On axial images, the distances between the tandem / central canal and the outer margins of hypo-echoic (dark) regions (TRUS based NMD's) can be utilized to guide the target contouring on the corresponding axial CT images. This methodology with use of TRUS is associated with a learning curve (approximately 10 -15 patients). Training module for the same are available on Brachtyterra (https://brachyterra.thinkific.com/).
3. CT Imaging with BT applicator in situ:

Standardized CT imaging protocol should be followed. CT imaging has to be performed with 1-1.5 ml/kg body weight iodine based intravenous contrast administration after utilizing a uniform bladder filling protocol for BT as defined in the Pre-BT MR protocol. During BT application, bladder is kept nearly empty with an indwelling catheter. At the time of CT Imaging, bladder cavity is instilled with 20 - 50 ml fluid (mixture of 1 ml of Sodium-meglumine diatrizoate 76%) contrast and 20-50 ml of normal saline) to achieve adequate contrast for outer wall contouring. A similar protocol using dilute contrast (10 - 15 ml) may be instilled into the recto-sigmoid, in addition to the rectal tube to assist in delineation of the rectum and sigmoid. CT imaging using ≤ 3 mm slice thickness should be performed, preferably include arterial/capillary phase or bolus tracking methods, to best define pelvic anatomy. Structures relevant to cervical cancer BT include primary tumor, cervical canal, cervix, vagina, uterine corpus, parametrium, pelvic vessels, uterine arteries, bladder, rectum and sigmoid. Training module for the same are available on Brachtyterra (https://brachyterra.thinkific.com/).

Applicator reconstruction and dose points for OARs:

Uncertainties of 4% (k=1) due to applicator reconstruction are assumed when reporting dose parameters for cervix brachytherapy. An appropriate step-by-step quality assurance program in each centre is compulsory as follows:

Step 1: The first step is to define source path (which is subsequent dwell positions of actual source inside applicator) in relation to applicator. This is usually defined during commissioning of applicators and after-loaders. The source path can be related to outer dimensions of an applicator/ marker wires or other indicators placed inside applicator. Autoradiographs are performed to visualize dwell positions. Commissioning procedure should result in determination of offsets (if any), drawings of essential dimensions or even applicator templates which can be integrated into treatment planning systems.

Step 2: Accuracy of applicator reconstruction depends on resolution of 3D image set. Appropriate imaging must be performed, either by reducing slice thickness, combining different image orientations (e.g. oblique orientations in transverse, sagittal and coronal) or using dedicated 3D sequences (e.g. isotropic voxel size). Each centre must ensure that applicator reconstruction can be performed with an uncertainty of < 2 mm. This includes overall deviation of planned dwell position to the finally realized dwell position on an anatomical situation as visualized on planning CT. This includes deviations due to source path definition (commissioning), equipment performance (constancy checks) and reconstruction process in treatment planning system.

Step 3: Direct reconstruction on CT or library plans may be an optimal solution for reducing uncertainties. Fusion of CT to Pre BT MRI / TRUS imaging is most often not helpful for applicator reconstruction, as fusion techniques have to be based on the already reconstructed applicator in both image modalities. Dose points for brachytherapy are defined directly on CT imaging with applicator in situ.

The following dose points should be defined directly in the 3D imaging study:

* Point 'A'
* ICRU bladder point
* ICRU recto-vaginal point Point A, recto-vaginal, and bladder reference points on CT as defined by ICRU 89 report must be strictly followed. Point A is a geometrical point in relation to applicator. A coordinate system is rotated and centred to have it aligned to applicator, with its origin in intrauterine applicator axis and the z=0 plane at the surface of the vaginal part of applicators. For defining recto-vaginal and bladder reference points, image orientation is essential. Both points are defined according to patient coordinate system - on anterior-posterior lines, which are strictly perpendicular to the longitudinal axis of the patient.

Contouring of target and organs at risk at BT:

Contouring of targets and OARs is performed for each BT applicator insertion / implant by contouring on axial CT images with BT applicator in situ, in a dedicated 3D brachytherapy dose- planning system according to GEC ESTRO ICRU 89 concept and IBS/ GEC-ESTRO/ ABS CT Recommendations.

No safety margins/ PTV margins are needed for internal movement ("tracking brachytherapy") since the applicator moves with the CTV. Although there are some uncertainties for setup (applicator reconstruction), these seem to be rather negligible, if systematic error can be kept below 2 mm and slice thickness below 5 mm (random error). In the present study it is therefore assumed that for BT no margins should be added to CTV, i.e. CTV = PTV.

Tumor targets and dose points:

• High risk target (CTV-THR): clinic-radiological macroscopic tumour extension at time of brachytherapy (GTVB) + whole cervix + presumed extra cervical tumour extension It should be noted that the CTV-THR target concept has been extrapolated from MR based target concepts. With mature clinical evidence (RetroEMBRACE, EMBRACE- I and many mono- institutional studies) for MR based target concept, CT based target concepts details are provided in the IBS GEC ESTRO ABS target recommendations. Clinical evaluation of CT based target concept is one of the main aims of the present study. Results obtained may then be used to further generate robust evidence and implement IGABT in regions where access to MR Imaging is limited or challenging.

CTV-THR-CT Contouring The CTV-THR-CT, can be defined and delineated based on the following information and documentation in various environments

* Clinical drawings / NMD's at diagnosis and at BT
* Imaging at diagnosis - CT or MR with documentation of NMD's
* Response categorization- Category I, II, or III.
* Pre-BT Imaging - Utilization of the NMD's on Pre-BT MR or representative TRUS images with tandem in place
* CT imaging with a defined protocol and BT applicator in situ is available.
* Defining width in the parametrial region utilizing NMD's (Clinical, Pre BT MR or TRUS), while thickness and height based on anatomical boundaries and the clinico-radiological environments.

For OARs the following organs and dose points should be defined:

Organs-at-risk:

OARs for routine CT based delineation include the rectum, bladder, sigmoid, bowel, while others like anal canal, vagina, urethra are recommended only when target volume and dose distribution are in close proximity. The definition of OARs follows anatomical boundaries and principles as detailed in ICRU 89.

For OAR volumes, organ outer walls have to be defined and delineated slice by slice using only one line as recommended by ICRU 89.

The assessment of small OAR volumes for brachytherapy planning and reporting (0.1 cm3 and 2 cm3) is applicable as recommended in ICRU 89 / GEC-ESTRO Recommendations II. For the rectum, a length of about 5 cm in cranio-caudal direction or longer related to vaginal sources needs to be delineated. Sigmoid colon, with specific focus on areas adjacent to uterus and target, should be clearly identified and contoured. Similarly, bowel loops have to be identified and areas (i.e., wall or organ volumes) near uterus need to be contoured with their entire circumference. The entire bladder including whole posterior, posterior-caudal (trigone), and posterior-cranial bladder wall should be delineated. For most of these parameters, in particular for 2 cm3 volume, a strong correlation has been demonstrated to clinical morbidity endpoints (eg cystitis, proctitis, fistula, vaginal stenosis, diarrhea.

* Bladder: The outer bladder wall is contoured.
* Rectum: The outer rectal wall is contoured from above the anal sphincter to the level of transition into the sigmoid
* Sigmoid: The outer sigmoid wall is to be contoured from the recto-sigmoid flexure to well above the parametria and the uterus (at least 2 cm)
* ICRU bladder point
* ICRU recto-vaginal point

Planning aims and dose prescription for IMPACT Based on the experience from MR-IGABT, all participating centres are encouraged to aim for a D90 dose of 85 to 95 Gy (EQD2) to CTV-THR without a major compromise in the OAR doses. However, there is no specific dose level recommended for target volume prescription in this study, as there is limited evidence for such recommendation using CT-IGABT. Therefore, every centre is encouraged to follow the specific institutional practice which reflects the clinical experience accumulated through implementation of MR-IGABT. Planning aims (soft constraints) and limits for prescribed dose (hard constraints) for treatment planning in Embrace II study should be used. In principle, the BT dose and fractionation scheduling is left to the discretion of individual participating institutions. However, recording and reporting process, must be uniform and in accordance with ICRU 89 reporting.

BT Planning and Dwell time optimisation:

The starting point in planning is usually a standard plan normalised to defined point A, which has been in use for a very long time for x-ray based BT in institutional tradition. It is recommended to follow this tradition in cases of only intracavitary as well as combined intracavitary/interstitial application geometries and adapt dose and volume according to specific individual needs of the clinical situation. It is not recommended to create a plan which is completely new, as this may imply uncertainties which may result in outcome, little predictable, the worst in significant adverse events.

STEP 1: Source loading which results in standardized pear shaped isodose distributions normalized to point A (sometimes named as standard plan) is usually achieved by certain loading patterns in the intrauterine and vaginal applicator parts. The balance of target dose coverage for defined volumes of target and OARs is achieved by optimization which is performed by optimising the implant geometry, the dwell time distribution and the fractionation.

STEP 2: The use of implant geometries with interstitial needles in addition to an intracavitary applicator is essential for unfavourable topography (either larger target volumes or unfavourable relation between target and OARs). It is assumed that at least 20 % of a representative cohort of cervical cancer cases needs such implant techniques to fulfil planning aims and prescription limits. The loading and dose contribution from the needles is added to the intracavitary dose distribution. This ensures that the dose levels and dose gradients around the implant geometry stay comparable to intracavitary plans and not interstitial plans, where each applicator has a similar weighting to avoid hot and cold spots in any areas not directly controlled via dose points or dose-volume relations. The contribution of TRAK resulting from the interstitial components to the overall TRAK varies on each situation, but is usually between 5-20 %.

The loading pattern and the dwell times are optimized in iterative steps until planning aims are fulfilled. Dwell time distribution can be optimised by using - (1) Manual dwell time or dwell weight optimization and/or (2) Graphical optimization ("dose shaping") combined with manual verification and adjustments for unnecessarily large deviations from typical pear shaped isodose with prescription to point A (also called standard loading pattern). Inverse planning tools are not recommended at present. It should only be used if individual centres perform reproducible and safe additional adaptations during or after inverse optimization process.

According to chapter 10.6.4 of the EMBRACE II protocol the dwell time optimization should not be solely based on dose and volume constraints. DVH constraints as suggested and used at present do not take into account high dose volumes within target and adjacent normal tissue. This applies for all organs where no recommendations for delineation have been developed so far (e.g. vagina, ureter, vessels, nerves or connective tissue in the pelvis). Therefore, to avoid any significant adverse clinical events specific attention is needed to ensure that dose distributions (especially for high dose volumes) are within the range and place of clinical experience collected so far and which seems to be achievable by not allowing for too large differences from traditional approaches. Especially the TRAK resulting from loading in the intrauterine applicator part, intravaginal applicator part and the interstitial needles should be monitored.

With increasing volume of CTV-THR-CT, the intravaginal applicator loading usually reaches a low plateau in TRAK and the intrauterine loading dominates the entire applied dose. Loading in the interstitial needles is lower compared to the intracavitary part and on average increases with target size. Only in case of extremely large CTV sizes, the interstitial component may reach TRAK values up to 50% of the entire TRAK, while it remains usually below 20% for the majority of cases.

Dose and volume recording and reporting All patients should receive both EBRT and BT. Summation of EBRT and BT doses will be performed by calculation of a biologically equivalent dose in 2 Gy per fraction (EQD2) using the linear-quadratic model with α/β of 10 Gy for tumour effects and α/β of 3 Gy for late normal tissue damage. The repair half time is assumed to be 1.5 hrs.

Recording and reporting follows the recommendations of ICRU/GEC ESTRO Report 89.

Reporting of dose and volume parameters for BT (from ICRU 89) CTV-THR-CT: Volume, D98, D90 Point A (only when intracavitary): Point dose Bladder: D2 cm³ Rectum: D2 cm³ Sigmoid: D2 cm³ and assessment of mobility Bowel: D2 cm³ and assessment of mobility ICRU recto-vaginal point: Point dose ICRU bladder point: Point dose TRAK: Total, needle, Vaginal

Quality Assurance:

Only approved departments and investigators can contribute patients to the protocol. It is the responsibility of the study coordinators to evaluate and approve participation. Approval requires a successful dummy run and an individual assessment of the performance of each participating centre. Online monitoring tools available at Medical University Vienna will be utilized. Centre based queries will be generated periodically for discussion and improve the quality of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Cancer of the uterine cervix considered suitable for curative treatment with definitive chemo radiotherapy including brachytherapy.
2. Biopsy showing invasive squamous-cell carcinoma or adenocarcinoma or adeno - squamous cell carcinoma of the uterine cervix.
3. FIGO (2018) stage IB2 to IVA
4. Willingness to participate by signing informed consent form.

Exclusion Criteria:

* Other previous or current primary malignancies except carcinoma in situ of the cervix.

  * Metastatic Inguinal Nodes not amenable to radical radiation therapy
  * Metastatic disease in para-aortic region beyond renal vessels
  * Not eligible for concurrent cisplatin chemotherapy (creatinine clearance < 50mg/ml/min)
  * Previous pelvic or abdominal radiotherapy.
  * Previous total or partial hysterectomy.
  * Patients receiving BT alone.
  * Patients receiving EBRT alone.
  * Patients receiving any form of neoadjuvant anti-neoplastic therapy prior to definitive treatment or adjuvant therapy
  * Active infection or severe medical condition which precludes radical chemoradiotherapy.
  * Pregnant or lactating or childbearing potential without adequate contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females diagnosed with cervical cancer
Study Population: The study will include approximately 1200 women with histologically confirmed, locally advanced cervical cancer (FIGO stages IB3-IVA) who are planned for curative chemoradiation followed by brachytherapy at the primary treating center. Participants will be recruited from multiple national and international centres equipped with CT-based brachytherapy facilities. All will undergo standardized treatment and follow-up as per study protocol, with imaging and outcome data submitted to a centralized database for quality assurance and analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Local control in relation to anatomical compartments and specific BT targets (CTV- THR) and morbidity related to OAR in the pelvis. | 36 & 60 Months
  Remission status (complete, partial, stable & progressive disease) should be evaluated 3 - 6 months after treatment by gynaecological examination and imaging wherever applicable. Regular follow-up including gynaecological examination with planned appointments 6, 9, 12, 18, 24, 30 and 36 months after treatment to be done & documented. In case of suspected recurrence, biopsy / fine needle aspiration cytology to confirm recurrences and appropriate imaging to be performed at the discretion of treating physician & Institutional protocol. Physician assessed morbidity will be scored prospectively with the Common Terminology Criteria for Adverse Events (both CTCAE V 5.0) on apriori selected, clinically relevant endpoints related to gastro-intestinal, genito-urinary, vaginal and several unspecific symptoms. Morbidity will be classified into early and late as per standard definition (early being within the first 90 days after completion of treatment).

SECONDARY OUTCOMES:
Regional control | 6, 9, 12, 18, 24, 30 and 36 months
  Remission status (complete, partial, stable & progressive disease) should be evaluated 3 - 6 months after treatment by gynaecological examination and imaging wherever applicable. Regular follow-up including gynaecological examination with planned appointments 6, 9, 12, 18, 24, 30 and 36 months after treatment to be done & documented. In case of suspected recurrence, biopsy / fine needle aspiration cytology to confirm recurrences and appropriate imaging to be performed at the discretion of treating physician & Institutional protocol.
Progression free survival | 6, 9, 12, 18, 24, 30 and 36 months
  Remission status (complete, partial, stable & progressive disease) should be evaluated 3 - 6 months after treatment by gynaecological examination and imaging wherever applicable. Regular follow-up including gynaecological examination with planned appointments 6, 9, 12, 18, 24, 30 and 36 months after treatment to be done & documented. In case of suspected recurrence, biopsy / fine needle aspiration cytology to confirm recurrences and appropriate imaging to be performed at the discretion of treating physician & Institutional protocol.
Overall survival | 6, 9, 12, 18, 24, 30 and 36 months
  Remission status (complete, partial, stable & progressive disease) should be evaluated 3 - 6 months after treatment by gynaecological examination and imaging wherever applicable. Regular follow-up including gynaecological examination with planned appointments 6, 9, 12, 18, 24, 30 and 36 months after treatment to be done & documented. In case of suspected recurrence, biopsy / fine needle aspiration cytology to confirm recurrences and appropriate imaging to be performed at the discretion of treating physician & Institutional protocol.
Morbidity | 6, 9, 12, 18, 24, 30 and 36 months
  Physician assessed morbidity will be scored prospectively with the Common Terminology Criteria for Adverse Events (both CTCAE V 5.0) on apriori selected, clinically relevant endpoints related to gastro-intestinal, genito-urinary, vaginal and several unspecific symptoms. Morbidity will be classified into early and late as per standard definition (early being within the first 90 days after completion of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Umesh Mahantshetty, MD, DNB, Principal Investigator — HOMI BHABHA CANCER HOSPITAL AND RESEARCH CENTRE
Locations (1):
- Homi Bhabha Cancer Hopsital & Research Centre, Visakhapatnam, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Haie-Meder C, Potter R, Van Limbergen E, Briot E, De Brabandere M, Dimopoulos J, Dumas I, Hellebust TP, Kirisits C, Lang S, Muschitz S, Nevinson J, Nulens A, Petrow P, Wachter-Gerstner N; Gynaecological (GYN) GEC-ESTRO Working Group. Recommendations from Gynaecological (GYN) GEC-ESTRO Working Group (I): concepts and terms in 3D image based 3D treatment planning in cervix cancer brachytherapy with emphasis on MRI assessment of GTV and CTV. Radiother Oncol. 2005 Mar;74(3):235-45. doi: 10.1016/j.radonc.2004.12.015. PMID 15763303
- [Result] Cibula D, Raspollini MR, Planchamp F, Centeno C, Chargari C, Felix A, Fischerova D, Jahnn-Kuch D, Joly F, Kohler C, Lax S, Lorusso D, Mahantshetty U, Mathevet P, Naik R, Nout RA, Oaknin A, Peccatori F, Persson J, Querleu D, Bernabe SR, Schmid MP, Stepanyan A, Svintsitskyi V, Tamussino K, Zapardiel I, Lindegaard J. ESGO/ESTRO/ESP Guidelines for the management of patients with cervical cancer - Update 2023. Virchows Arch. 2023 Jun;482(6):935-966. doi: 10.1007/s00428-023-03552-3. Epub 2023 May 5. PMID 37145263
- [Result] Miriyala R, Sreelakshmi KK, Chiriki K, Hajare R, Vadgaonkar R, Nachu S, Grover S, Mahantshetty U. GPP06 Presentation Time: 9: 45 AM: Early Clinical Outcomes of Cervical Cancer Treated with CT Based Image Guided Adaptive Brachytherapy Using IBS-GEC ESTRO-ABS Recommendations. Brachytherapy. 2024 Nov 1;23(6):S19.
- [Result] Mahantshetty U, Naga Ch P, Khadanga CR, Gudi S, Chopra S, Gurram L, Jamema S, Ghadi Y, Shrivastava S. A Prospective Comparison of Computed Tomography with Transrectal Ultrasonography Assistance and Magnetic Resonance Imaging-Based Target-Volume Definition During Image Guided Adaptive Brachytherapy for Cervical Cancers. Int J Radiat Oncol Biol Phys. 2018 Dec 1;102(5):1448-1456. doi: 10.1016/j.ijrobp.2018.05.080. Epub 2018 Jun 7. PMID 30146092
- [Result] Potter R, Tanderup K, Kirisits C, de Leeuw A, Kirchheiner K, Nout R, Tan LT, Haie-Meder C, Mahantshetty U, Segedin B, Hoskin P, Bruheim K, Rai B, Huang F, Van Limbergen E, Schmid M, Nesvacil N, Sturdza A, Fokdal L, Jensen NBK, Georg D, Assenholt M, Seppenwoolde Y, Nomden C, Fortin I, Chopra S, van der Heide U, Rumpold T, Lindegaard JC, Jurgenliemk-Schulz I; EMBRACE Collaborative Group. The EMBRACE II study: The outcome and prospect of two decades of evolution within the GEC-ESTRO GYN working group and the EMBRACE studies. Clin Transl Radiat Oncol. 2018 Jan 11;9:48-60. doi: 10.1016/j.ctro.2018.01.001. eCollection 2018 Feb. PMID 29594251
- [Result] Mahantshetty U, Poetter R, Beriwal S, Grover S, Lavanya G, Rai B, Petric P, Tanderup K, Carvalho H, Hegazy N, Mohamed S, Ohno T, Amornwichet N. IBS-GEC ESTRO-ABS recommendations for CT based contouring in image guided adaptive brachytherapy for cervical cancer. Radiother Oncol. 2021 Jul;160:273-284. doi: 10.1016/j.radonc.2021.05.010. Epub 2021 May 18. PMID 34019918
- [Result] Potter R, Tanderup K, Schmid MP, Jurgenliemk-Schulz I, Haie-Meder C, Fokdal LU, Sturdza AE, Hoskin P, Mahantshetty U, Segedin B, Bruheim K, Huang F, Rai B, Cooper R, van der Steen-Banasik E, Van Limbergen E, Pieters BR, Tan LT, Nout RA, De Leeuw AAC, Ristl R, Petric P, Nesvacil N, Kirchheiner K, Kirisits C, Lindegaard JC; EMBRACE Collaborative Group. MRI-guided adaptive brachytherapy in locally advanced cervical cancer (EMBRACE-I): a multicentre prospective cohort study. Lancet Oncol. 2021 Apr;22(4):538-547. doi: 10.1016/S1470-2045(20)30753-1. PMID 33794207
- See also: Improving cervical cancer care through personalized radiation therapy PROMISE, IMPACT, and REWIND studies for image-guided adaptive brachytherapy. — https://www.embrace-triplet.org